CLINICAL TRIAL: NCT00230243
Title: A Retrospective Study to Establish an Historical Database on the Efficacy of Standard Antifungal Therapy in Patients With Invasive Fungal Infections
Brief Title: Historical Control Study of Refractory IFI or Patients Intolerant to Standard Antifungal Therapy in Patients With Invasive Fungal Infections (Study P02387)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P02387
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Infection, Invasive Fungal
Keywords: Aspergillosis; CandidiasisMucormycosis; FusariosisCryptococcosis; Endemic Fungal infections; Phaeohyphomycosis
MeSH Terms: conditions — Invasive Fungal Infections; Aspergillosis; Phaeohyphomycosis

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This retrospective study is designed to provide a consistent method of screening and collecting data on patients who will serve as controls for a comparison of the efficacy of the available antifungal therapies used as salvage treatments for patients with refractory IFI or for patients with refractory IFI or for patients with IFI who are intolerant to standard antifungal therapies.

DETAILED DESCRIPTION:
The current clinical trial is designed to provide historicals controls comparable to the P00041 study population, that is, a) patients with invasive fungal infections which are refractory or resistant to standard antifungal therapies or b) patients who have developed intolerance to standard antifungal therapy. This clinical trial also serves to allow collection of historical data regarding the efficacy of available antifungal therapies against a variety of invasive fungal infections which although serious and life-threatening are sufficiently rare so that they cannot be studied in a controlled, randomized clinical trial.

This trial will be conducted primarily at the investigative sites that enrolled subjects into P00041 and/or investigators who are members of the Mycosis Study Group.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any race greater than or equal to 13 years of age
* Treatment for an IFI between April 30, 1996 and April 30, 2001 at one of the centers participating in P00041 or at other non-P00041 centers
* A diagnosis of proven or probable IFI based on MSG/EORTC criteria
* Refractory IFI or intolerence to standard therapy

The date of diagnosis of an IFI will be the earliest date on which one or more of the following diagnostic procedures used to establish the diagnosis was performed:

* Fungal culture, histopathology, bronchoscopy, and autopsy report
* X-Rays, CT scan, MRI, ultrasound, and bone scan
* Serology

Exclusion Criteria:

1. Female subject who was pregnant or nursing at the time IFI was diagnosed
2. Hepatic function tests: ALT or AST greater than 10 times the upper limit of normal at the time IFI was diagnosed
3. Enrollment in P00041 for treatment of the IFI
4. Patient with sarcoidosis, aspergilloma, or allergic bronchopulmonary aspergillosis
5. Patients with chronic invasive aspergillosis (chronic necrotizing pulmonary aspergillosis)
6. Patients with diagnosis of CMV pneumonia
7. Patients with a diagnosis of pulmonary tuberculosis
8. Death within 72 hours of the start of antifungal therapy
9. Patients on artificial ventilation, who were not extubated within 24 hours of commencing standard antifungal therapy

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330
Dates: Start 1997-03; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html